CLINICAL TRIAL: NCT05374135
Title: Effect of Dexamethasone on Fetal Heart Rate Variables In Case Of Imminent Preterm Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ereny Wagih Youssif, Ereny wagih youssif, Assiut University
Other Study IDs: Dexamethasone effect on FHR
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Fetal Heart Rate or Rhythm Abnormality Affecting Fetus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Effect of dexamethasone on fetal heart rate variability in case of preterm labour: prospective cohort study

DETAILED DESCRIPTION:
prospective cohort study on Effect of dexamethasone on fetal heart rate variability in case of preterm labour

ELIGIBILITY:
Inclusion Criteria:

* Preterm labor

Exclusion Criteria:

* Twins

Ages: 15 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Changes in fetal heart rate variability in relation to dexamethasone administration | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Kh Al-Hussini, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt